CLINICAL TRIAL: NCT05884918
Title: Risk Factors and Frequency of Intraoperative Hypotension in High-risk Patients Undergoing Surgery: A Multicenter Observational Prospective Study
Brief Title: Intraoperative Hypotension in High-risk Patients Undergoing Surgery
Acronym: IRIoHYP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mazovia Regional Hospital in Siedlce (Other)
Responsible Party: Principal Investigator, Jolanta Cylwik, Principal Investigator, Mazovia Regional Hospital in Siedlce
Other Study IDs: 1/2023
Record Dates: First submitted 2023-05-12; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia; Hypotension on Induction; Perioperative Injury; Perioperative Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this observational study is to investigate the risk factors for intraoperative hypotension and identify the underlying pathomechanisms leading to it, both during the period after general anesthesia induction and throughout its course.

The main questions it aims to answer are:

* how frequent is intraoperative hypotension
* what are the underlying pathomechanism causing it The study is including patients who have been identified as having a high risk of perioperative complications (ASA3 or ASA4). Patients included in the study undergo advanced hemodynamic monitoring during the procedure. Anesthesia induction, maintenance, and termination are conducted by an anesthesiologist in accordance with current medical knowledge, and the planned experiment does not in any way influence the course of action.

Investigators will analyse medical documentation, including the patient's medical history, anesthesia records, and hemodynamic parameter data obtained from the hemodynamic monitor (an Excel file containing comprehensive data related to specific cardiovascular parameters) to describe the incidence of intraoperative hypotension and answer key questions in accordance with the designed study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Capability of providing informed consent by the patient.
* Planned surgeries.
* Surgeries other than thoracic, cardiac, or obstetric procedures.
* ASA (American Society of Anesthesiologists) physical status classification of 3 or 4, indicating high risk.
* Patients at high risk of postoperative complications.
* Preoperative qualification for advanced hemodynamic monitoring.
* Access to complete preoperative health status data.
* Access to complete data regarding the course of anesthesia and hemodynamic parameters obtained from the hemodynamic monitoring platform.
* Initiation of hemodynamic monitoring prior to general anesthesia induction.

Exclusion Criteria:

* Age <18 years old.
* Cardiac surgeries.
* Thoracic surgeries.
* Obstetric procedures.
* Inability of the patient to provide informed consent.
* ASA physical status classification of 1, 2, or 5, indicating low or moderate risk.
* Urgent and emergent surgeries.
* Lack of complete preoperative health status data.
* Lack of complete data regarding the course of anesthesia.
* Inability to initiate hemodynamic monitoring prior to general anesthesia induction.
* Interruption in hemodynamic monitoring lasting longer than 5 minutes (lack of parameter values in the obtained hemodynamic monitor file).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age: > 18 years old. Gender: Women and men. Preoperative qualification for advanced hemodynamic monitoring based on the estimated high risk of postoperative complications.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension (IOH) | Intraoperative
  Incidence of IOH due to the general anesthesia
Risk factors of IOH. | Perioperative
  Rate of specific clinical and demographical parameters associated with IOH

SECONDARY OUTCOMES:
Development of a risk scale for IOH (MAP < 65mmHg) based on the identified risk factors in the study. | Perioperative
  Combination of the most significant risk factors of IOH into risk scale.
Determination of indications for intraoperative extended hemodynamic monitoring. | Perioperative
  List of pre-operative clinical factors indicating elevated risk of peri-operative complications
Assessment of the incidence, duration, and depth of hypotension as a complication of general anesthesia at each stage of anesthesia. | Perioperative
  List of specific parameters related to IOH.
Evaluation of the relationship between the depth and duration of hypotensive episodes and the occurrence of postoperative complications within 30 days of the surgical procedure. | Perioperative to 30 days after surgery
  List of clinical factors associated with IOH impacting clinical adverse events during 30 days follow up.
Analysis of the anesthesiologist's management approach in the event of hypotensive episodes or hypotension risks and an attempt to establish an optimal management strategy for its occurrence. | Perioperative
  List of routine actions triggered by the IOH in the anesthesiological management.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Cylwik, PhD, Principal Investigator — Mazovian Regional Hospital in Siedlce, Poland
Locations (1):
- Mazovian Regional Hospital, Siedlce, Mazovian, Poland